CLINICAL TRIAL: NCT05511779
Title: Phase II, Open-label, Randomized, Multiple Ascending Dose Confirmation of the Safety and Tolerability of Brincidofovir in Subjects With BK Virus Infection (Viremia) After Kidney Transplantation (BASTION)
Brief Title: Study to Confirm of the Safety and Tolerability of Brincidofovir in Subjects With BK Virus Infection (Viremia) After Kidney Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to delays in enrollment
Sponsor: SymBio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BCV-BN01
Record Dates: First submitted 2022-08-16; First posted 2022-08-23 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: BK Virus Infection; Nephropathy; Kidney Transplantation
Keywords: BK Virus; Nephropathy; Kidney transplantation
MeSH Terms: conditions — Kidney Diseases | interventions — brincidofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose Escalation Phase: Cohort 1: BCV 0.3 mg/kg BIW (Experimental): BCV: 0.3 mg/kg administered as a continuous IV infusion over 2 hours on Day1 and Day4 for 8 weeks (up to a maximum of 14 weeks).
  Interventions: Drug: Brincidofovir
- Dose Escalation Phase: Cohort 2: BCV 0.4 mg/kg BIW (Experimental): BCV: 0.4 mg/kg administered as a continuous IV infusion over 2 hours on Day1 and Day4 for 8 weeks (up to a maximum of 14 weeks).
  Interventions: Drug: Brincidofovir
- Expansion Phase: BCV Recommended dosage regimen in the Dose Escalation Phase (Experimental): BCV: Recommended dosage administered as a continuous IV infusion over 2 hours on Day1 and Day4 for 8 weeks (up to a maximum of 14 weeks).
  Interventions: Drug: Brincidofovir

INTERVENTIONS:
Drug: Brincidofovir — BCV 0.3 mg/kg BIW or 0.4 mg/kg BIW administered as a continuous IV infusion over 2 hours
  Other Names: SyB V-1901; BCV

SUMMARY:
This is a Phase II, multicenter, open-label, randomized, standard of care (SOC) controlled, multiple ascending dose study to assess the safety and tolerability of IV Brincidofovir (BCV) in subjects with BKV infection after kidney transplantation. The study will be conducted at multiple study sites in several countries including Australia and Japan. Subjects who meet eligibility criteria will be enrolled in the study and will be randomized and assigned to BCV or SOC (defined as use of the same immunosuppressant administered during prescreening) before receipt of the first dose of study drug in both the Dose Escalation Phase and the Expansion Phase.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years of age at the time of signing the informed consent at screening.
* Kidney transplant recipient. "BK viral load increase and ≥ 3.6 log IU/mL" at 2 weeks post immunosuppression reduction or "BK viral load does not decrease by ≥ 0.3 log IU/mL" at 4 weeks post immunosuppression reduction during prescreening.

(Note: Immunosuppressant reduction needs to be continued during the screening period).

* eGFR ≥ 30 mL/min.
* Subjects under immunosuppression with tacrolimus, MMF/Myfortic, and/or corticosteroid.

Exclusion Criteria:

* Subjects who weigh ≥ 120 kg.
* National Institutes of Health/NCI CTCAE Grade 2 or higher diarrhea (ie, increase of ≥ 4 stools per day over usual pretransplant stool output) within 7 days before Day 1.
* Poor clinical prognosis, including active malignancy or use of vasopressors other than low dose (eg, ≤ 5 μg/kg/min) dopamine for renal perfusion within 7 days before Day 1.
* Use of renal replacement therapy within 7 days before Day 1.
* History of intolerance to cidofovir or related compounds (ie, other nucleotide derivatives [adefovir or tenofovir])

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2023-04-13 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | from the time of administration of the first dose of study drug through the follow-up visit(up to 14 weeks (treatment period) and 30 days (follow-up period))
  * Incidence of TEAEs of the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade 3 severity and serious adverse events
  * Incidence of treatment-related TEAEs
  * Incidence of adverse events (AEs) requiring permanent discontinuation of BCV
  * Absolute and changes over time in safety laboratory parameters (ie, hematology, blood chemistry, and urinalysis)
Antiviral Effects | From baseline to follow-up visit(up to 14 weeks (treatment period) and 30 days (follow-up period))
  Change from baseline in BK viral load in plasma measured through follow-up for each subject. Change from baseline in BK viral load in urine measured through follow-up for each subject. Peak BK viral load in plasma from Week 2 Day 1 through follow-up for each subject. Time-averaged area under the viremia-time curve for BK viral load in plasma from baseline through follow-up for each subject.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wojciechowski D, Kotton CN. BK Nephropathy in the Modern Era: What Have We Learned? Kidney360. 2025 Dec 1;6(12):2257-2262. doi: 10.34067/KID.0000000967. Epub 2025 Aug 19. PMID 40828617
- [Derived] Wajih Z, Karpe KM, Walters GD. Interventions for BK virus infection in kidney transplant recipients. Cochrane Database Syst Rev. 2024 Oct 9;10(10):CD013344. doi: 10.1002/14651858.CD013344.pub2. PMID 39382091